CLINICAL TRIAL: NCT01644461
Title: A Prospective, Multicentric, Open Label, Bio-Interventional, Phase I/II Pilot Study To Evaluate The Safety And Efficacy Of Autologous Human Platelet Lysate (HPL) For Treatment of Facial Wrinkles (Nasolabial Folds)
Brief Title: A Study to Determine Safety & Efficacy of Autologous Human Platelet Lysate (HPL) in Facial Wrinkles(Nasolabial Folds)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kasiak Research Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KRPL/HPL-FR/11-12/002B
Record Dates: First submitted 2012-07-17; First posted 2012-07-19 (Estimated); Last update posted 2012-07-25 (Estimated); Status verified 2012-07

CONDITIONS: Facial Wrinkles (Nasolabial Folds)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Study Group (Other): All subjects will receive a single injection of Autologous Human Platelet Lysate in the nasolabial region
  Interventions: Other: Autologous Human Platelet Lysate

INTERVENTIONS:
Other: Autologous Human Platelet Lysate — All subjects will receive a single injection of Autologous Human Platelet Lysate in the nasolabial region

SUMMARY:
This is a multicentre, open label, pilot study to evaluate safety and efficacy of Autologous Human Platelet Lysate (HPL) in subjects with Facial Wrinkles (Nasolabial Folds). The study is being conducted at 2 centers in India. The primary endpoints are Improvement in Wrinkle Severity Rating Scale ( WSRS ) as per ATLAS photographic grading at rest and on full smile and Global Aesthetic Improvement Scale (GAIS). The secondary endpoints are improvement in photographic assessment, Physician's assessment scores, Patient's assessment scores form enrollment to end of study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects (male and female), aged 18 to 40 years (both inclusive).
* Subjects willing to refrain from any other treatment for Nasolabial Folds.
* Subjects who are willing to give informed consent and adhere to the study protocol.

Exclusion Criteria:

* Subjects receiving any aesthetic facial therapy 6 months prior to enrolment e.g. Botox, Fillers etc
* Subjects with history of Connective tissue disease
* Subjects with autoimmune diseases
* Subjects unwilling to or unable to comply with the study protocol.
* Subjects taking concomitant therapy that might interfere with the study results in the investigator's opinion or participating in another trial in the past 30days

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-04; Primary Completion 2012-10 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
Wrinkle Severity Rating Scale as per ATLAS photographic grading at rest & on full smile | Day 0, End of Study - 3 months

SECONDARY OUTCOMES:
Global Aesthetic Improvement Scale | Day 0, End of study - Month 3

OTHER OUTCOMES:
Photographic assessments | Day 0, Month 1, Month 2, End of study - Month 3
Physician's assessment scores | End of Study - 3 months
Patient's assessment scores | End of Study - 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Rachita Dhurat, Dr., Principal Investigator — Dr Rachita's Skin, Trichology & Aesthetic Centre; Geetanjali Shetty, Dr., Principal Investigator — Kapadia Multispeciality Hospital
Locations (1):
- Kasiak Research Pvt Ltd, Thane, Maharashtra, India